CLINICAL TRIAL: NCT02429479
Title: Preparing Family Caregivers of Very Ill Patients for End-of-Life Decision Making
Brief Title: Preparing Family Caregivers to Make Medical Decisions for Their Loved Ones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Benjamin H. Levi, Co-PI, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 37476; 1R01NR012757-01A1 (NIH)
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Last update posted 2024-01-26 (Actual); Status verified 2021-08

CONDITIONS: Neoplasms; Heart Failure; Kidney Diseases; Lung Diseases
Keywords: Advance Care Planning; Living Will; Family Caregiver; Advance Directive; Surrogate Decision Maker; Proxy; Self-Efficacy
MeSH Terms: conditions — Neoplasms; Heart Failure; Kidney Diseases; Lung Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard ACP/Patient Alone (Active Comparator): Patients (without their family caregiver) complete a standard living will form online.
  Interventions: Behavioral: Standard advance care planning
- Decision Aid/Patient Alone (Experimental): Patients (without their family caregiver) complete Making Your Wishes Known, an online decision aid for advance care planning.
  Interventions: Behavioral: Making Your Wishes Known
- Standard ACP/Together (Active Comparator): Patients and their family caregiver together complete a standard living will form online.
  Interventions: Behavioral: Standard advance care planning
- Decision Aid/Together (Experimental): Patients and their family caregiver together complete Making Your Wishes Known, an online decision aid for advance care planning.
  Interventions: Behavioral: Making Your Wishes Known

INTERVENTIONS:
Behavioral: Making Your Wishes Known — Making Your Wishes Known provides tailored education, values clarification exercises, and a sophisticated decision aid that translates an individual's goals and preferences into a specific medical plan that can be implemented by a healthcare team.
  Arms: Decision Aid/Patient Alone; Decision Aid/Together
Behavioral: Standard advance care planning — This is a online simple living will form.
  Arms: Standard ACP/Patient Alone; Standard ACP/Together

SUMMARY:
The overarching goal of the project is to improve the process and experience of surrogate decision-making by family caregivers. Since feeling unprepared to make surrogate decisions is a major contributor to caregiver stress, the primary outcome is caregiver self-efficacy --i.e., caregivers' assessment of how well prepared they feel to serve effectively as a surrogate decision-maker. Through follow-on Renewal funding, we are now also qualitatively examining family caregivers' experience with surrogate decision-making.

DETAILED DESCRIPTION:
The long-term goal is to help family caregivers of seriously ill patients be better prepared to serve as surrogate decision-makers when their loved ones can no longer make medical decisions for themselves. Research shows that family caregivers find surrogate decision-making highly stressful and emotionally burdensome, in part because they feel unprepared for surrogate decision-making. To date, no studies have determined which advance care planning (ACP) process best prepares caregivers for this role. The investigators' prior work shows that a computer-based decision aid can help patients make more informed decisions and communicate their wishes more effectively. The investigators now propose to determine if family caregivers of patients with life-threatening illnesses are better prepared for surrogate decision-making: 1) when they engage in a structured ACP process together with patients; and 2) when they use this online decision aid for ACP. This will be accomplished via a randomized, controlled trial with a 2 x 2 factorial design comprising 4 groups: Standard ACP/Patient Alone (Group 1), Decision Aid/Patient Alone (Group 2), Standard ACP/Patients and Caregivers Together (Group 3), and Decision Aid/Patients and Caregivers Together (Group 4).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Diagnosis of kidney disease (e.g. chronic kidney disease, end stage renal disease ) OR advanced cancer (Stage IV disease or having an estimated survival of <2 years) OR severe heart failure (e.g. New York Heart Assoc. Class III or Class IV) OR severe lung disease (e.g. Stage III or Stage IV COPD by modified GOLD Spirometric Classification, Idiopathic Pulmonary Fibrosis).
3. Able to read and understand English at an 8th grade level (word 26 on either blue or tan version of the WRAT-3 reading subtest)
4. Neuro-cognitively able to engage in ACP (Mini Mental State Exam (MMSE) score >23)
5. No active suicidal ideations (i.e., score of 0 or 1 on item 9 of the BDI-II).

Exclusion Criteria:

* Failure on any of the above inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Self-efficacy | 6 weeks
  Family caregiver self-efficacy is measured using a validated questionnaire to determine if they feel better prepared to serve as surrogates for their loved one.

SECONDARY OUTCOMES:
Accuracy of medical decisions | 6 weeks
  Family caregiver responses to treatment decisions hypothetical clinical vignettes will be compared to the decisions for the same vignettes made by their loved one. Each vignette has 6-8 associated treatment decisions; the family caregiver's response for each item will be compared with the loved one's (i.e., patient's) response, and a total concordance (i.e., number of items for which there is agreement) will be calculated.
Family caregivers' stress associated with actual (i.e., real-life) surrogate decision-making | 1-2 years
  Using validated instruments and semi-structured interviews, family caregivers who have made a major medical decision on behalf of their loved one will report their level of distress, decisional conflict, satisfaction with decision, and experience with surrogate decision-making.
Family caregiver knowledge | 6 weeks - 2 years
  Family caregivers will complete a questionnaire that assess their knowledge of surrogate responsibilities and end-of-life medical conditions and treatments
Depth of communication | 2 years
  Family Caregivers are interviewed about the depth of communication with their loved one (frequency, content, helpfulness of discussions) regarding advance care planning issues.
Satisfaction with advance care planning | 1st study visit
  Participants who complete the advance care planning interventions fill out an evaluation of the intervention using a 16-item questionnaire. This instrument comprises:
  Twelve 5-point Likert-style questions on how the program presented various kinds of information; helped the user clarify values, choose a spokesperson, etc.; and helped the user document or be prepared communicate their wishes to others.
  Three 10-point Likert-style questions on user overall satisfaction, with the advance directive created by the intervention, and the amount of information provided.
  One open-ended item asking how the intervention was helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin H Levi, MD PhD, Principal Investigator — Penn State Milton S. Hershey Medical Center / Penn State College of Medicine; Michael J Green, MD MS, Principal Investigator — Penn State Milton S. Hershey Medical Center / Penn State College of Medicine
Locations (2):
- United States (2):
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Penn State Milton S. Hershey Medical Center / Penn State College of Medicine, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
We will present our findings at conferences and in peer-reviewed publications, and will share our study protocol, consent forms, measures, and statistical plan with other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: July 1, 2023 - June 30, 2026
Access Criteria: Researchers who provide a methodologically sound proposal/request for these data.

REFERENCES:
- [Derived] Thiede E, Levi BH, Lipnick D, Johnson R, Seo La I, Lehman EB, Smith T, Wiegand D, Green M, Van Scoy LJ. Effect of Advance Care Planning on Surrogate Decision Makers' Preparedness for Decision Making: Results of a Mixed-Methods Randomized Controlled Trial. J Palliat Med. 2021 Jul;24(7):982-993. doi: 10.1089/jpm.2020.0238. Epub 2020 Dec 29. PMID 33373538
- [Derived] Lipnick D, Green M, Thiede E, Smith TJ, Lehman EB, Johnson R, La IS, Wiegand D, Levi BH, Van Scoy LJ. Surrogate Decision Maker Stress in Advance Care Planning Conversations: A Mixed-Methods Analysis From a Randomized Controlled Trial. J Pain Symptom Manage. 2020 Dec;60(6):1117-1126. doi: 10.1016/j.jpainsymman.2020.07.001. Epub 2020 Jul 6. PMID 32645452
- [Derived] Foy AJ, Levi BH, Van Scoy LJ, Bucher A, Dimmock A, Green MJ. Patient Preference to Accept Medical Treatment Is Associated with Spokesperson Agreement. Ann Am Thorac Soc. 2019 Apr;16(4):518-521. doi: 10.1513/AnnalsATS.201806-428RL. No abstract available. PMID 30714833